CLINICAL TRIAL: NCT04286477
Title: The Immune System in End Stage Chronic Kidney Disease (CKD) Patients - Comparison Among Different Modalities of Renal Replacement Therapy (RRT)
Brief Title: The Immune System in End Stage CKD Patients - Comparison Among Different Modalities of RRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Ioannina (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Evangelia Ntounousi, Assistant Professor, University of Ioannina
Other Study IDs: RESCOMUOI82758
Record Dates: First submitted 2020-02-13; First posted 2020-02-27 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: Peritoneal Dialysis; Hemodiafiltration; Expanded Hemodialysis; Monocytes subpopulations; Regulatory T cells; Natural Killer cells; Lymphocytes

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 15 conventional hemodialysis patients: 15 patients undergoing hemodialysis with high-flux dialyzer
- 15 patients undergoing online-hemodiafiltration: 15 patients undergoing conventional hemodialysis with high-flux dialyzer will be allocated to online-hemodiafiltration with the same dialyzer
- 15 patients undergoing expanded hemodialysis with MCO dialyzer: 15 hemodialysis patients undergoing hemodialysis with a high-flux dialyzer will be allocated to HDx with an MCO dialyzers (THERANOVA dialyzer, Baxter International Inc. (NYSE: BAX))
- 15 patients undergoing peritoneal dialysis: 15 patients undergoing peritoneal dialysis

SUMMARY:
The evaluation and assessment of the influence of the different modalities of renal replacement therapy (RRT), including peritoneal dialysis (PD), conventional hemodialysis with high flux dialyzers, hemodiafiltration (HDF) and expanded hemodialysis (HDx) with Medium Cut Off (MCO) dialyzers on the levels of the cell subsets of the innate and acquired immune system as well as the investigation of the possible role of these cells as prognostic indices of morbidity and mortality in patients with end-stage Chronic Kidney Disease (CKD) undergoing different modalities of RRT.

DETAILED DESCRIPTION:
The sustained inflammatory state in CKD is of complex pathogenesis and is believed to be in part attributable to the augmented activation of innate immune system cell subsets. The activation of the innate immune system plays an essential role within all the spectrum of cardiovascular disease in CKD, including accelerated atherosclerosis, left ventricular hypertrophy and heart failure. However, the intricate immunological mechanisms involved in the pathogenesis of CKD-associated cardiovascular disease remain to be clarified.The hemodialysis procedure itself is associated with an increased inflammatory burden. Considering the fact that middle molecules lie at the crossroads of chronic inflammation and immune dysregulation, oxidative stress as well as cardiovascular morbidity of CKD, efforts have focused on improving the clearance of larger middle molecules in dialysis. Hemodiafiltration is considered to further improve the clearance of larger toxins by utilizing large-volume ultrafiltration, also known as convection. HDF compared with standard hemodialysis, may have beneficial effects with regard to micro-inflammation, as indicated by lower levels of inflammatory markers, C-reactive protein (CRP), and Interleukin 6 (IL-6). However, evidence from large outcome trials comparing HDF to hemodialysis is controversial The introduction of the newest generation of highly selective and permeable MCO, which have an increasingly porous membrane but with tightened distribution of pore sizes, is associated with increased removal of large middle-molecules up to a molecular weight of 45,000 Dalton (Da). On the other hand safety concerns regarding MCO membranes such as albumin loss and back filtration of endotoxins have proven to be inconsistent by clinical studies run so far. Accordingly the clinical benefits of MCO membranes with regard to patient outcomes,chronic inflammation, immune dysregulation, atherosclerosis or structural heart disease, remains to be evaluated by future clinical studies. Until now there are no data regarding the effects of expanded hemodialysis on immune cell subsets or comparative studies regarding the influence of the currently available methods of RRT on immune cell subsets with expanded hemodialysis. Whether expanded hemodialysis with MCO membranes is associated with "improved" patterns of immune cell subsets with regard to chronic micro-inflammation as compared to the currently available methods, including HDF, and whether this translates into improved clinical outcomes remains to be elucidated, this being the aim of our study.

30 patients undergoing conventional hemodialysis and 15 patients undergoing PD will be enrolled in the study. The study will be designed in two arms - the cross-sectional arm and the prospective arm during which patients will be under follow-up for 12 months.

The cross-sectional study:

Immune cell subtypes will be measured at baseline in all patients. In patients undergoing hemodialysis, measurements will be performed in the midweek dialysis session and for PD patients during a programmed visit at the PD unit.

Regarding patients undergoing conventional hemodialysis:

* 15 of those undergoing conventional hemodialysis with high-flux dialyzers will be allocated to online-HDF with the same dialyzer and 15 hemodialysis patients undergoing hemodialysis with a high-flux dialyzer will be allocated to HDx with MCO dialyzers (THERANOVA dialyzer, Baxter International Inc. (NYSE: BAX)), for 12 consecutive weeks. Immune cell subtypes will be measured in the midweek dialysis session of the 12th week.
* subsequently both groups will be allocated to conventional hemodialysis with the same dialyzer as baseline for another 4 weeks as a wash-out phase and thereafter they will be crossed over to online-HDF and HDx with the THERANOVA dialyzer for another 12 week period. Immune cell subtypes will be measured in the midweek dialysis session of the 28th week.

Thereafter, patients will proceed with the hemodialysis modality, which they were allocated to during the last 12 weeks of the study and immune cell subtypes will be measured 20 weeks later. The overall duration of the study will be 48 weeks. Immune cell subtypes will be measured in the midweek dialysis session of the 48th week. Regarding peritoneal dialysis, immune cell subtypes will be measured at baseline and at 48 weeks.

The evaluation of the immune cells subtypes will be done by flow-cytometry of peripheral blood. The following cell types will be measured:

1. CD14++C16-, CD14+CD16+, CD 14+CD16++ subpopulations of monocytes
2. Natural Killers (NK cells
3. CD4+ lymphocytes and CD8+ lymphocytes
4. CD 4+CD25+ Τ regulatory lymphocytes (Tregs) (CD = Cluster of Differentiation)

Demographic data and anthropometric data, major cardiovascular risk factors, the cause of end-stage CKD, co-morbidities and medical treatment shall be recorded for all patients at baseline.

A cardiovascular workout will take place. All hemodialysis patients will undergo at baseline, week 12 and week 28:

* echocardiographic evaluation with estimation of classical and novel echocardiographic parameters of systolic and diastolic left ventricular function,
* ABP (Ambulatory Blood Pressure) monitoring
* Carotid Doppler for the estimation of intima-media thickness (IMT)
* Lung ultrasound for the assessment of lung comets

PD patients shall undergo the same diagnostic procedures as hemodialysis patients at baseline and at week 48.

Additional routine blood test examinations shall be performed monthly, including complete blood count and biochemical blood tests including glucose, blood urea nitrogen (BUN), creatinine, potassium, sodium, calcium, phosphate, serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT), creatine kinase (CPK), gamma-glutamyltransferase (γGT), alkaline phosphatase (ALP), proteins and albumin, immunoglobulins, lipid panel - total cholesterol, triglycerides, low-density lipoproteins (LDL), high-density lipoproteins (HDL) - uric acid, iron, total iron binding capacity (TIBC), ferritin, parathyroid hormone (PTH), vitamin D, CRP, erythrocyte sedimentation rate (ESR), fibrinogen.

Dialysis adequacy (monthly KT/V, urea reduction rate (URR) in hemodialysis patients and quarterly KT/V, residual renal function as well as peritoneal function testing in PD patients shall be regularly monitored according to international guidelines.

Nutritional parameters and hydration status shall be evaluated at baseline, at week 12 and at week 28 in hemodialysis patients and quarterly in PD patients.

During the prospective arm of the study (12 months) data regarding technique failure, infections, hospitalizations for any cause and major cardiovascular events (acute coronary syndrome, cerebrovascular accident, heart failure, peripheral vascular disease, sudden cardiac death) and death from any cause will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* adult patients between 18 and <90 years
* CKD G5 (glomerular filtration rate (GFR) <15 ml/min/1.73m2)
* conventional hemodialysis treatment thrice weekly for at least three months via permanent vascular access
* patients undergoing PD for at least three months.

Exclusion Criteria:

* presence of infection
* active malignancy
* liver cirrhosis
* inflammatory bowel disease
* active autoimmune disease
* decompensated heart failure (New York Heart Association (NYHA) IV
* occurence of a major cardiovascular event within less that three months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients undergoing RRT in the Hemodialysis and PD Unit of the Nephrology Department of the University Hospital of Ioannina. Patients will be informed with regard to the study and they will provide written informed consent before enrollment. The study will be approved by the Ethics Committee of the University Hospital of Ioannina.
  Accordingly, adult patients between 18 and 90 years and CKD G5 (GFR < 15ml/min/ 1.73m2) requiring conventional hemodialysis treatment thrice weekly, since at least three months via a permanent vascular access (fistula, graft or a tunneled central venous catheter) and patients undergoing PD (continuous ambulatory peritoneal dialysis (CAPD) or Automated peritoneal dialysis (APD)) for at least three months.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2018-11-07 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the peripheral blood levels of the cell subsets of the innate and acquired immune system in patients with end-stage CKD transitioning from hemodialysis to hemodiafiltration or expanded hemodialysis. | 1st-12th week
  Immune cell subtypes (CD14++CD16- monocytes, CD14++CD16+ monocytes, CD 14+CD16+ monocytes, NK cells, CD4+ lymphocytes, CD8+ lymphocytes and Tregs) will be measured by flow cytometry at baseline in patients undergoing hemodialysis in the midweek dialysis session. 15 of patients undergoing conventional hemodialysis will be allocated to online-HDF with the same dialyzer and 15 conventional hemodialysis patients will be allocated to HDx with an MCO dialyzer (THERANOVA dialyzer, Baxter International Inc. (NYSE: BAX)), for 12 weeks. Immune cell subtypes will be measured in the 12th week.
Comparison of the peripheral blood levels of the cell subsets of the innate and acquired immune system in patients with end-stage CKD undergoing hemodiafiltration versus expanded hemodialysis. | 12th-28th
  Patients allocated to online-HDF and patients allocated to HDx with an MCO dialyzer (THERANOVA dialyzer, Baxter International Inc. (NYSE: BAX)), will be allocated to conventional hemodialysis for 4 weeks as a wash-out phase and then they will be crossed over to online-HDF and HDx with THERANOVA dialyzer for 12 weeks. Immune cell subtypes (CD14++CD16- monocytes, CD14++CD16+ monocytes, CD 14+CD16+ monocytes, NK cells, CD4+ lymphocytes, CD8+ lymphocytes and Tregs)will be measured by flow cytometry in the 28th week.
Comparison between the peripheral blood levels of the cell subsets of the innate and acquired immune system in patients with end-stage CKD undergoing hemodialysis, hemodiafiltration, expanded hemodialysis and peritoneal dialysis. | 12-28th
  Immune cell subtypes (CD14++CD16- monocytes, CD14++CD16+ monocytes, CD 14+CD16+ monocytes, NK cells, CD4+ lymphocytes, CD8+ lymphocytes and Tregs)will be measured in 15 PD patients during a programmed visit at the PD unit.

SECONDARY OUTCOMES:
Correlation between peripheral blood levels of the cell subsets of the innate and acquired immune system with dialysis adequacy, adequacy of fluid control, nutritional indices, and inflammatory markers. | 1st - 48th week
  Correlations will be made between peripheral blood levels of CD14++CD16- monocytes, CD14++CD16+ monocytes, CD 14+CD16+ monocytes, NK cells, CD4+ lymphocytes, CD8+ lymphocytes and Tregs (at all time points measured as described in primary otcome) as assessed with flow cytometry with dialysis adequacy (KT/V, URR, residual renal function), adequacy of fluid control (dry body weight, body composition monitoring (BCM), lung ultrasound), nutritional indices (serum albumin, normalized protein catabolic rate (nPCR) and inflammatory markers (CRP, serum ferritin, IL-6, tumor necrosis factor α (TNFα, growth and differentiation factor 15 (GDF15), galectin3, interleukin 1 receptor-like 1 also known as ST2 etc.).
Correlation between peripheral blood levels of the cell subsets of the innate and acquired immune system with established cardiovascular disease, atherosclerosis markers, indicesof systolic and diastolic cardiac function and occurrence of infections. | 1st - 48th week
  A correlation will be sought between peripheral blood levels of CD14++CD16- monocytes, CD14++CD16+ monocytes, CD 14+CD16+ monocytes, NK cells, CD4+ lymphocytes, CD8+ lymphocytes with presence of established cardiovascular disease (heart failure, ischemic heart disease), markers of atherosclerosis (IMT), with indices of systolic and diastolic cardiac function (left ventricular ejection fraction (LVEF), E and A wave, mitral annular plane systolic excursion (MAPSE) septal and lateral, deceleration time, left atrium dimensions, pulmonary artery systolic pressure, inferior vena cava diameter) and finally with occurrence of infections.
Prognostic indices of morbidity (hospitalizations, cardiovascular events, infections) and mortality (due to any cause or cardiovascular mortality). | 24 months
  The prospective part of the study will be the investigation of the possible role of the evaluated cell subsets of the innate and acquired immune system (monocyte subsets, NK cells, CD4 and CD8 lymphocytes and T regs) as prognostic indices of morbidity (hospitalizations, cardiovascular events, infections) and mortality (due to any cause or cardiovascular mortality).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece

REFERENCES:
- [Background] Heine GH, Ulrich C, Seibert E, Seiler S, Marell J, Reichart B, Krause M, Schlitt A, Kohler H, Girndt M. CD14(++)CD16+ monocytes but not total monocyte numbers predict cardiovascular events in dialysis patients. Kidney Int. 2008 Mar;73(5):622-9. doi: 10.1038/sj.ki.5002744. Epub 2007 Dec 26. PMID 18160960
- [Background] Vacher-Coponat H, Brunet C, Lyonnet L, Bonnet E, Loundou A, Sampol J, Moal V, Dussol B, Brunet P, Berland Y, Dignat-George F, Paul P. Natural killer cell alterations correlate with loss of renal function and dialysis duration in uraemic patients. Nephrol Dial Transplant. 2008 Apr;23(4):1406-14. doi: 10.1093/ndt/gfm596. Epub 2007 Nov 20. PMID 18029366
- [Background] Caprara C, Kinsey GR, Corradi V, Xin W, Ma JZ, Scalzotto E, Martino FK, Okusa MD, Nalesso F, Ferrari F, Rosner M, Ronco C. The Influence of Hemodialysis on T Regulatory Cells: A Meta-Analysis and Systematic Review. Blood Purif. 2016;42(4):307-313. doi: 10.1159/000449242. Epub 2016 Oct 1. PMID 27694753
- [Background] Kim HW, Yang HN, Kim MG, Choi HM, Jo SK, Cho WY, Kim HK. Microinflammation in hemodialysis patients is associated with increased CD14CD16(+) pro-inflammatory monocytes: possible modification by on-line hemodiafiltration. Blood Purif. 2011;31(4):281-8. doi: 10.1159/000321889. Epub 2011 Jan 14. PMID 21242682
- [Background] Wolley M, Jardine M, Hutchison CA. Exploring the Clinical Relevance of Providing Increased Removal of Large Middle Molecules. Clin J Am Soc Nephrol. 2018 May 7;13(5):805-814. doi: 10.2215/CJN.10110917. Epub 2018 Mar 5. PMID 29507008